CLINICAL TRIAL: NCT03753971
Title: Early Sleep Apnea Termination Using Sound Stimulation
Acronym: ESAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Raphael Heinzer (Other)
Responsible Party: Sponsor-Investigator, Raphael Heinzer, Professor, University of Lausanne Hospitals
Organization: University of Lausanne Hospitals (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19121997; 2018-02033 (Other: Swissethics)
Record Dates: First submitted 2018-11-08; First posted 2018-11-27 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apneas with and without intervention (Experimental): Each patient will be his own control.
  Interventions: Other: Sound stimulation

INTERVENTIONS:
Other: Sound stimulation — Short sound stimulations will be emitted through a head band during sleep apneas

SUMMARY:
Current evidence suggest that sleep apnea-associated oxygen desaturations may induce cardiovascular morbidities in the long term, whereas arousals associated with sleep apneas seem to induce mainly transient nocturnal hypertension. Reducing the occurrence and the magnitude of sleep apnea-associated oxygen desaturations could therefore have a beneficial effect on sleep apnea-associated comobidities. Since sleep apneas usually end with an arousal allowing pharyngeal muscles reactivation, a treatment option could consist of generating an early short awakening to anticipate apnea termination and decrease the risk of oxygen desaturation. The aim of this study is thus to determine if an early sleep apnea termination through the emission of a sound can achieve lower oxygen desaturations compared with "untreated" sleep apneas.

DETAILED DESCRIPTION:
The aim of the study is to determine the effect of short sound stimulations on sleep apnea associated desaturations

20 OSA subjects will be recruited and studied with polysomnography and a head band allowing to emit short sound stimulations during sleep. the study will take nplace at the Center for investigation and research in sleep (CIRS)

The magnitude of oxygen desaturations following apnea with and without sound stimulations will be compared. The effects of different types of sound stimulations on the magnitude of cortical and autonomic reactions will also be studied as well as the patients' subjective perception of the sounds.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Able to give informed consent as documented by signature
* Apnea / hypopnea index > 30 / h (severe)
* Obstructive Apnea Index > 15 / h
* Mean amplitude of desaturations (during diagnostic night) ≥ 5%

Exclusion Criteria:

* Perception deafness
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc.,
* Professional drivers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-01-16 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Differences in sleep apnea associted oxygen desaturations | During the polysomnography night
  Differences in the magnitude of blood oxygen desaturation between treated and untreated sleep apnea events (in % of SaO2)

SECONDARY OUTCOMES:
Duration of the apnea (seconds) | During the polysomnography night
  Duration of breathing cessation assessed by nasal cannula (in seconds)
Percentage of sound stimulations associated with cortical and subcortical arousals (%) | During the polysomnography night
  Each arousal will be assessed using the polysomnography EEG
Percentage of sound stimulations associated with autonomic arousals (%) | During the polysomnography night
  Autonomic arousals will be assessed by pulse wave amplitude variations
Magnitude of autonomic reactions (% of pulse wave amplitude drop) | During the polysomnography night
  Magnitude (% of baseline) of pulse wave amplitude drop following different types of sound stimulations
Duration of EEG arousals (in seconds) | During the polysomnography night
  Duration (in seconds) of EEG arousals following different types of sound stimulations
Magnitude of autonomic reactions (duration of pulse wave amplitude drop) | During the polysomnography night
  Duration of pulse wave amplitude drop following different types of sound stimulations (in seconds)

OTHER OUTCOMES:
Patients' perception of the sounds emitted during sleep (visual analog scale 0-10) | Morning after the polysomnography night
  Perception of the sound stimulations (number per night)
Patients' tolerance to the sounds (visual analog scale 0-10) | Morning after the polysomnography
  VAS scale reflecting the annoyance associted with the sounds emitted during their sleep

CONTACTS AND LOCATIONS:
Overall Officials: Raphael Heinzer, Pr., Study Director — Centre d'investigation et de recherche sur le sommeil (CHUV)
Locations (1):
- Adrien Waeber, Jouxtens-Mézery, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Waeber A, Arnal PJ, Lecciso G, Albir D, Mignot E, Heinzer R. Acoustic stimulation time-locked to the beginning of sleep apnea events reduces oxygen desaturations: a pilot-study. Sleep Med. 2021 Feb;78:38-42. doi: 10.1016/j.sleep.2020.12.006. Epub 2020 Dec 11. PMID 33383395